CLINICAL TRIAL: NCT06164678
Title: Vaping Cessation Using the Ottawa Model for Smoking Cessation Among E-Cigarette Users: A Pilot RCT
Brief Title: Vaping Cessation Using the Ottawa Model for Smoking Cessation Among E-Cigarette Users
Acronym: VC-OMSC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230670-01H
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Smoking; Vaping
MeSH Terms: conditions — Tobacco Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1
Who Masked: Investigator, Outcomes Assessor
Masking Description: A blinded member of the research team will complete all follow-up assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ottawa Model for Smoking Cessation (Experimental): The OMSC group will receive counselling and pharmacotherapy if they choose (specifically NRT) with follow-up calls to support medication titration. Participants will be provided with quit cards, which are pre-loaded with $300 worth of funds that can only be used by the assigned study participant to purchase NRT (if they choose).
  For those in the intervention group, the study counsellor who is a trained Nicotine Addiction Treatment Specialist (NATS) will facilitate follow-up, monitor NRT use, and advise participants to titrate NRT dose as required based on their minimum daily nicotine intake. These counselling calls will be conducted at day 3, 7, 14, 21, 30, 60, 90, and 180 as is standard in OMSC for people who smoke and are interested in quitting. A diary will also be provided to the participants to track their usage.
  Interventions: Behavioral: OMSC
- Usual Care (No Intervention): The usual care group will receive the initial counselling session but no further follow-up or NRT. They will be able to self-initiate a follow-up call if they choose. Participants will not be excluded if they choose to initiate NRT on their own at their own expense.

INTERVENTIONS:
Behavioral: OMSC — The OMSC program uses a counselling approach to assist clients with tobacco cessation. If required, nicotine replacement therapy may be offered.
  Arms: Ottawa Model for Smoking Cessation

SUMMARY:
This study aims to determine if a standardized approach including counselling and Nicotine Replacement Therapy (NRT) can help e-cigarette users quit vaping. Current e-cigarette users will be randomly assigned to either to counselling and NRT or counselling only group. Self-reported rates of vaping cessation will be measured throughout the year in both groups. The use of e-cigarettes has grown substantially among non-smokers, particularly among youth and young adults. These devices deliver high levels of nicotine, far greater than is possible with conventional cigarettes. Currently, they are not approved for smoking cessation or any purpose by Health Canada. Nonetheless, there is some evidence that e-cigarettes may be of assistance in smoking cessation. Conversely, there is evidence that using cigarettes and e-cigarettes together may result in increased cigarette consumption. E-cigarette use among youth also serves as a gateway to regular use of conventional cigarettes. Clinicians and patients are seeking guidance on vaping cessation. However, to date, there are no strong evidence-based interventions to support e-cigarette users in quitting. NRT is approved for smoking cessation by Health Canada. However, it is not approved for vaping cessation and thus its use to support e-cigarette users to quit by managing their nicotine withdrawal is considered "off-label". This represents a significant gap and opportunity, which this project will address.

The study hypothesizes that the OMSC approach, which includes the use of nicotine replacement therapy, will result in higher rates of vaping cessation compared to usual care.

Participants will all complete an initial counselling session to discuss vaping cessation and receive tips to help achieve cessation. They will all be asked to track their smoking/vaping behaviour and the amount of tobacco in their e-cigarette for 7 days. After 7 days, all participants will be randomly put into one of two groups (either the intervention or control group). They will have follow-up assessments with the research team at 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age or older
* Ontario resident
* Ability to speak English or French
* Regular use of e-cigarette (vaping at least once per week for the past four weeks)

Exclusion Criteria:

* Cognitive impairment or acute psychiatric illness that would alter their ability to participate
* Being institutionalized at a retirement home, nursing home or long-term care facility
* Participating in another smoking or vaping cessation program
* Allergy or intolerance to NRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Vaping Cessation | baseline to 3 months
  7-day point prevalence of vaping cessation measured at 3-months.

SECONDARY OUTCOMES:
Continuous Abstinence | 1-day, 7-day, 1-month, 3-month, 6-month, and 12-month from baseline date
  Continuous abstinence rates at 1-day, 7-day, 1-month, 3-month, 6-month, and 12-month follow up.
Successful cessation | 12 month assessment
  Self-reported cessation will be measured by a self-administered salivary cotinine test.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mir, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No